CLINICAL TRIAL: NCT04229667
Title: Optimising a Community-based Model for Case Identification, Monitoring, and Prevention of Hypertension and Diabetes Among Syrian Refugees in Jordan
Brief Title: Community Models for Hypertension and Diabetes Care for Refugees
Status: Terminated | Type: Observational
Why Stopped: As a result of COVID-19, the intervention design changed and an RCT was no longer an appropriate study design for evaluation.
Sponsor: International Rescue Committee (Other)
Collaborators: University of Southern California (Other); Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: H 1.00.020
Record Dates: First submitted 2019-10-24; First posted 2020-01-18 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Hypertension; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Comorbidities and Coexisting Conditions
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Improved Community Health Volunteer (CHV) program — Multi-modal intervention targeting intensive household monitoring of "high-needs" patients using monthly visits to measure blood pressure and blood sugar, adherence to treatments and compliance with clinics visits, and motivational interviewing to facilitate behavior change and psychosocial support.

SUMMARY:
The project will investigate and improve a community health worker (CHW) based model for non-communicable disease (NCD) care in a humanitarian emergency.

DETAILED DESCRIPTION:
Guidelines for public health approaches for non-communicable disease (NCD) in crises are not well developed. More broadly, NCD management in developing countries focuses on care at the health facility level without a community health worker focus (CHW), which may facilitate continuous care and monitoring.

Since the arrival of refugees from Syria in 2012, the International Rescue Committee (IRC) has provided primary health care, mobile outreach, and community-based empowerment programs for those in need in the northern governorates of Mafraq and Ramtha. The IRC runs health clinics, mobile medical teams, and community health volunteer (CHV) networks to provide care for refugees and Jordanians living in poverty.

This stepped-wedge observational study will follow the implementation of an improved CHV program which focuses on the monitoring of 'high-needs' patients in their households for complications, severe disease, and to avoid interruptions to treatment adherence. The stepped-wedge design will be undertaken to benefit from the phased rollout of the improved CHV intervention over a year-long period. The intervention will be scaled to 20 CHV-neighborhoods across Mafraq and Ramtha.

Primary objectives:

* To evaluate the impact of an improved CHV program that targets high-needs hypertension and diabetes patients on:
* Compliance with routine clinic visits.
* Adherence to medications (self-reported).
* Adherence behaviours (self-reported).
* Disease control outcomes (blood pressure control for hypertension patients; blood sugar control for diabetes patients).

Secondary objectives:

* To document the operations of the improved CHV program in terms of key operational indicators and health indicators.
* To produce lessons learned to improve the CHV program.

Study outcomes:

* Evidence of the effectiveness of the improved CHV strategy on clinic visit compliance, adherence, and patient outcomes.
* Improved guidance for developing and implementing an integrated model of primary care and community health worker networks in crises.

ELIGIBILITY:
Inclusion Criteria:

Adult (≥18 years of age) with clinically-diagnosed hypertension OR type II diabetes AND;

1. Poor adherence, defined as:

   - Missed ≥2 appointments in the past six months AND/OR;
2. Poor disease control:

   Hypertension: Blood pressure >160/90 (EHS/ESC Grade II/III) with or without therapy, on their last measurement in clinic AND/OR; Evidence of hypertensive end organ damage including ischemic heart disease, left ventricular hypertrophy on ECG, eGFR < 60, hypertensive retinopathy, heart failure, myocardial infarction AND/OR; Type II diabetes: HbA1C is >8.5% OR random blood glucose >200 mg/dL with or without insulin/pill therapy AND/OR; Patient has comorbidity and/or evidence of diabetic end organ damage, including ischemic heart disease, left ventricular hypertrophy on ECG, eGFR < 60, retinopathy, heart failure, myocardial infarction, poorly healing wounds (e.g., diabetic foot), amputation, blindness and eye problems.
3. Comorbid diabetes and hypertension:
4. Disabled (house-bound)
5. Type I diabetes (insulin-dependent): all adult cases of insulin-dependent diabetes (likely type I diabetes), due to the nature of treatment interruption which causes rapid decompensations.

Exclusion Criteria:

* Pregnancy
* Hospitalization for the majority of the study period
* Patients who leave the study neighborhood or repatriate to Syria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years), Syrian refugee or vulnerable Jordanian patients with type 1 or type 2 diabetes mellitus and/or hypertension and considered to have "high-needs", living in the IRC-clinic catchment areas of Ramtha and Mafraq, Jordan
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of diabetes patients at intake (defined as random blood sugar >= 200 mg/dL at intake) demonstrating a change in random blood sugar (mmHg) | Every two months, through study completion (4 to 12 months depending on group)
  As measured by point-of-care glucometer
Proportion of hypertension patients at intake (defined as blood pressure >=140/90 mmHg at intake) demonstrating a change in systolic blood pressure (mmHg) | Every two months, through study completion (4 to 12 months depending on group)
  As measured by electronic blood pressure monitor during household visit
Proportion of patients demonstrating a change in self-reported medication adherence behaviors | Every two months, through study completion (4 to 12 months depending on group)
  As measured by response to questions on adherence behaviors. This measure uses the Center for Adherence Support Evaluation (CASE) Adherence Index, wherein higher values on a scale of 1 to 6 indicate worse outcomes.
Proportion of patients demonstrating a change in self-reported medication adherence actions (5-day) | Every two months, through study completion (4 to 12 months depending on group)
  As measured the number of days during the last 5 days in which medication was not taken (during household visit)
Proportion of patients demonstrating a change in self-reported medication adherence actions (30-day) | Every two months, through study completion (4 to 12 months depending on group)
  As measured the number of days during the last 30 days in which medication was not taken (during household visit)

SECONDARY OUTCOMES:
Proportion of hypertension patients at intake (defined as blood pressure >=140/90 mmHg at intake) demonstrating a change in diastolic blood pressure (mmHg) | Every two months, through study completion (4 to 12 months depending on group)
  As measured by electronic blood pressure monitor during household visit
Proportion of patients demonstrating a change in disease control (defined as blood pressure <140/90 mmHg; <150/90 for patients aged ≥80 years), among patients with hypertension at intake (defined as blood pressure >=140/90 mmHg at intake) | Every two months, through study completion (4 to 12 months depending on group)
  As measured by electronic blood pressure monitor using three measurements during household visit
Proportion of patients demonstrating a change in disease control (defined as random blood sugar <200 mg/dL mmHg), among patients with diabetes at intake (defined as random blood sugar >=200 mg/dL at intake) | Every two months, through study completion (4 to 12 months depending on group)
  As measured with glucometer during household visit

CONTACTS AND LOCATIONS:
Locations (1):
- International Rescue Committee, New York, New York, United States